CLINICAL TRIAL: NCT06501833
Title: Efficacy of FIFA 11+ Kids Injury Prevention Program on Soccer-specific Skills Among Young Soccer Players- A Randomized Controlled Trial
Brief Title: Efficacy of FIFA 11+ Kids Injury Prevention Program on Soccer-specific Skills Among Young Soccer Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Shibili Nuhmani, Assistant professor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-PGS-2023-03-254
Record Dates: First submitted 2024-06-26; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Healthy Young Soccer Players

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA 11+ kids program group (Experimental)
  Interventions: Other: FIFA 11+ KIDS PROGRAM
- Regular training group (Active Comparator)
  Interventions: Other: REGULAR TRAINING

INTERVENTIONS:
Other: FIFA 11+ KIDS PROGRAM — The experimental group will perform eight weeks of FIFA 11+ kids program (3/week).
  Arms: FIFA 11+ kids program group
Other: REGULAR TRAINING — The control group will be continuing their regular training
  Arms: Regular training group

SUMMARY:
Background: Soccer is a prevalent sport worldwide; most soccer players are under 18. Soccer has benefits for your health, but there is also a chance that you could get injuries occasionally. High injury rates have been observed in both adult and young players, which has prompted the development of various preventive measures. FIFA recently introduced the FIFA 11+ Kids program for children under 14 to prevent soccer injuries and enhance kids' performance. To date, no studies have been done to determine whether adding the FIFA 11 + kids program for young players under 14 will enhance soccer-specific skills.

Objective: To investigate the efficacy of FIFA 11+ Kids on soccer-specific skills among young soccer players.

Methods: Thirty six young soccer players (aged 7-13) will be assigned randomly to the following groups: the control group (n =18) and the FIFA 11+ Kids program (n = 18). The experimental group will perform eight weeks of FIFA 11+ kids program (3/week). The control group will be instructed to continue their regular training . Three soccer specific skills tests : the Slalom dribble test, Harre circuit test, and Loughborough soccer passing test, will be done before and after eight weeks of training.

Statistical analysis: IBM SPSS software (version 20) will be used for all statistical analyses. Data will be summarized in terms of mean and SD. Normality is checked with the Shapiro-Wilk test and homogeneity with Levene's tests. If the data are normally distributed, a paired t-test will be used for within-group difference comparison, and an independent t-test will be used for between-group comparison. If the data are not normally distributed, the Wilcoxon-Signed rank and Mann-Whitney U tests will be used.

ELIGIBILITY:
The inclusion criteria are

1. Healthy male young soccer players between the ages of 7-13 (al Attar et al., 2022).
2. Playing experience of at least one year.
3. Participating in a training session at least three times per week (Teixeira et al., 2021).
4. Participating in training at least 4.5 hours a week.

The exclusion criteria:

1. Upper or lower limb injuries require medical attention within the last six months (al Attar et al., 2022).
2. Any systemic disease, cardiovascular, neurological disorders, or surgery may affect the measurement and participation as reported by the participants (al-Attar et al., 2022).
3. Any medication which may affect the training or measurement as reported by the participants.
4. Any biomechanical abnormalities as reported by the participants.
5. Missed two consecutive training sessions or three separate ones (Mirwald et al., 2002).
6. Missing one of the testing sessions (Mirwald et al., 2002).

   -

Ages: 7 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Slalom dribble test | pre and immediately post intervention
Harre circuit test | pre and immediately post intervention
Loughborough soccer passing test | pre and immediately post intervention